CLINICAL TRIAL: NCT06654947
Title: A Single-arm, Open-label, Prospective Clinical Study of Surufatinib Combined With Immunotherapy and Chemotherapy for Unresectable or Metastatic Biliary Tract Cancer.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST-BTC-001
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-10

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Experimental (Experimental)
  Interventions: Drug: Surufatinib+Toripalimab+GEMOX

INTERVENTIONS:
Drug: Surufatinib+Toripalimab+GEMOX — Surufatinib (200mg，qd，Q3W）；Toripalimab(240mg IV d1, Q3W)；GEMOX：Gemcitabine: 1000 mg/m2, IV，d1，d8，Q3W，Oxaliplatin：100mg/m2,ivgtt，d1，Q3W）

SUMMARY:
This is a single-arm, open-label, prospective clinical study aimed at observing and evaluating the efficacy and safety of surufatinib combined with immunotherapy and chemotherapy in the treatment of unresectable or metastatic biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully comprehended this study and voluntarily signed the Informed Consent Form;
2. Age ≥ 18 years;
3. Inoperable or metastatic biliary tract carcinoma confirmed by histopathology or cytology;
4. Hepatic function classified as Child-Pugh Class A (scores 5-6) or Class B with favorable prognosis (score ≤7) (refer to Appendix 3);
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (refer to Appendix 1);
6. Anticipated survival ≥ 12 weeks;
7. At least one measurable lesion according to RECIST 1.1 criteria (refer to Appendix 2);
8. Essentially normal function of major organs and bone marrow:

   1. Complete blood count: WBC ≥ 4.0 × 10^9/L, neutrophils ≥ 1.5 × 10^9/L, platelets ≥ 100 × 10^9/L, hemoglobin ≥ 90 g/L;
   2. Prothrombin time expressed as International Normalized Ratio (INR) ≤1.5 × upper limit of normal (ULN), and activated partial thromboplastin time (APTT) ≤1.5 × ULN;
   3. Hepatic function tests: Total bilirubin ≤ 1.5 × ULN; without liver metastasis, ALT/AST/ALP ≤ 2.5 × ULN; with liver metastasis, ALT/AST/ALP ≤ 5 × ULN;
   4. Renal function tests: Serum creatinine ≤ 1.5 × ULN, and creatinine clearance (CCr) ≥ 60 mL/min (refer to Appendix 6);
   5. Cardiac function within normal limits, with left ventricular ejection fraction (LVEF) ≥ 50% as determined by two-dimensional echocardiography.
9. Male or female patients of reproductive potential voluntarily agree to use effective contraception during the study and for six months following the final administration of study medication, such as dual-barrier methods, condoms, oral or injectable contraceptives, intrauterine devices, etc. All female patients will be considered to have reproductive potential unless they have undergone spontaneous menopause, surgically-induced menopause, or have had a hysterectomy, bilateral salpingectomy, or ovarian irradiation with radioisotopes.

Exclusion Criteria:

1. Patients who relapsed within 6 months after previous immunosuppressive therapy;
2. Clinically symptomatic central nervous system metastases and/or carcinomatous meningitis;
3. Biliary obstruction that, in the investigator's judgment, has not resolved or requires anti-infective treatment within 14 days prior to the first study drug administration despite clinical intervention;
4. History of liver transplantation;
5. Active autoimmune disease or immunodeficiency;
6. Any surgery or invasive treatment or procedure (excluding venous catheterization, puncture drainage, etc.) within 4 weeks prior to study enrollment;
7. Uncontrolled hypertension not managed with medication, defined as: systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100 mmHg;
8. Urinalysis indicating proteinuria ≥2+ and, with a 24-hour urine protein quantification >1.0g;
9. Current presence of any disease or condition affecting drug absorption, or the patient's inability to orally ingest sorafenib;
10. Current active gastric and duodenal ulcers, ulcerative colitis, or other gastrointestinal diseases, or active bleeding from an unresected tumor, or other conditions deemed likely to cause gastrointestinal bleeding or perforation by the investigator;
11. Active bleeding or severe bleeding tendency;
12. Significant clinical cardiovascular disease, including but not limited to acute myocardial infarction within 6 months prior to enrollment, severe/unstable angina, or coronary artery bypass grafting; New York Heart Association (NYHA) classification > grade 2 for congestive heart failure; ventricular arrhythmias requiring drug therapy; electrocardiogram (ECG) showing QTc interval ≥480 milliseconds;
13. Active or uncontrolled severe infection (≥Grade 2 infection by CTC AE);
14. Known human immunodeficiency virus (HIV) infection; known clinically significant liver disease history, including viral hepatitis [known carriers of hepatitis B virus (HBV) must exclude active HBV infection, i.e., HBV DNA positive (>1×10^4 copies/mL or >2000 IU/mL); known hepatitis C virus (HCV) infection and HCV RNA positive (>1×10^3 copies/mL), or other types of hepatitis, cirrhosis];
15. Unresolved toxicities higher than Grade 1 by CTCAE from any previous anticancer treatment, excluding alopecia, lymphocytopenia, and ≤Grade 2 neurotoxicity caused by oxaliplatin (excluding well-controlled immune-related thyroiditis and pituitary inflammation with hormone replacement therapy);
16. Pregnant (positive pregnancy test before medication) or breastfeeding women;
17. Any other disease, clinically significant metabolic abnormalities, physical examination abnormalities, or laboratory test abnormalities that, in the investigator's judgment, reasonably suspect the patient has a certain disease or condition unsuitable for the use of the study medication (such as epilepsy requiring treatment), or will affect the interpretation of the study results, or place the patient at high risk.
18. Received strong inducers or inhibitors of cytochrome P450 (CYP) 3A within 2 weeks or 5 half-lives (whichever is longer) prior to the first dose of study medication;
19. A history of malignant tumors other than the current tumor within 5 years prior to screening, except for those with negligible risk of metastasis or death (e.g., overall 5-year survival rate >90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin cancer, localized prostate cancer, carcinoma in situ of the breast, or stage I uterine cancer; The investigator deems that the patient has other factors that may affect the study results or lead to premature termination of this study, such as alcohol abuse, drug abuse, other serious diseases (including mental illnesses) requiring concurrent treatment, significant laboratory test abnormalities, accompanied by family or social factors that will affect patient safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  Tumor assessment will be performed using radiography method every 6 weeks, until the occurrence of progressive disease (PD), using RECIST v 1.1

SECONDARY OUTCOMES:
Objective response rate (ORR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  Tumor assessment will be performed using radiography method every 6 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
Overall survival (OS） | from randomization until death due to any cause, assessed up to 3 year
  Tumor assessment will be performed using radiography method every 6 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
Disease control rate (DCR） | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  Tumor assessment will be performed using radiography method every 6 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
Safety and tolerance evaluated by incidence, severity and outcomes of AEs | from first dose to 30 days post the last dose
  Safety and tolerance will be evaluated by incidence, severity and outcomes of AEs and categorized by severity in accordance with the NCI CTC AE Version 5.0

IPD SHARING:
Plan to Share IPD: No